CLINICAL TRIAL: NCT01498029
Title: A Randomised Clinical Trial Comparing a Novel Single-stage Autologous Cartilage Implantation System to Conventional Microfracture for Repair of Articular Cartilage Defects in the Knee
Brief Title: Knee Articular Cartilage Repair: Cartilage Autograft Implantation System Versus Conventional Microfracture
Acronym: CAIS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CART/ 5 April 2011
Record Dates: First submitted 2011-12-07; First posted 2011-12-23 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2011-12

CONDITIONS: Other Articular Cartilage Disorders; Osteochondritis Dissecans
Keywords: Cartilage, Articular
MeSH Terms: conditions — Osteochondritis Dissecans | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Randomized to Microfracture (Active Comparator): This group of patients who have been randomised to receive microfracture procedure will be the control group for this study
  Interventions: Procedure: Microfracture
- Randomized to CAIS (Experimental): This group of patients who have been randomised to receive the CAIS procedure will be the experimental group for this study
  Interventions: Device: Cartilage Autograft Implantation System (CAIS)

INTERVENTIONS:
Procedure: Microfracture — The microfracture procedure is a standard method for treatment of cartilage damage in which the surgeon will clean the site of your cartilage damage and then will make several small holes in your bone to stimulate your bone marrow with the intention to repair the damaged area with new cartilage tissue
  Other Names: Knee; Cartilage; Cartilage Repair
  Arms: Randomized to Microfracture
Device: Cartilage Autograft Implantation System (CAIS) — The Cartilage Autograft Implantation System (CAIS) is a kit of devices that utilizes morselized autologous hyaline cartilage harvested arthroscopically, affixed onto a synthetic, resorbable implant using a fibrin sealant and implanted in a single surgical procedure. The system is designed as a surgical treatment of damaged knee cartilage using the subject's own healthy cartilage obtained from a non-weight or low weight-bearing region.
  Other Names: Knee; Cartilage; Cartilage Repair
  Arms: Randomized to CAIS

SUMMARY:
The Cartilage Autograft Implantation System (CAIS) is a single-stage procedure in which cartilage is harvested from non-critical regions of articular cartilage, but then immediately morcellated and loaded onto a polymer membrane-scaffold, which is subsequently used to fill the chondral defect. The autograft-membrane composite is fixed to the defect with a biodegradable staple.

The investigators aim to evaluate this new technique through a pilot clinical trial involving 36 patients randomized into microfracture and CAIS treatment arms (randomisation ratio 1:2), with a minimum follow-up of 1 year, using both clinical and radiological (magnetic resonance imaging) outcomes. If the results of this pilot trial are successful, the investigators plan to expand the study by recruiting more patients to achieve a suitably-powered trial.

Primary hypothesis 1: That functional scores will increase by at least 0.5 SD over pre-operative values, by 1 year following the CAIS procedure

Primary hypothesis 2: That articular cartilage height will have a sustained increase of at least 2 mm at 1 year following the CAIS procedure

Primary hypothesis 3: That functional scores in the CAIS group will be equivalent or superior to those in the microfracture group

DETAILED DESCRIPTION:
Articular cartilage has limited potential for regeneration, and full-thickness cartilage defects in the knee are frequently symptomatic and debilitating. If left untreated, such injuries may progress to generalized osteoarthritis. The management of these injuries remains unsatisfactory despite intense research activity, and the clinical and social impact of this problem is growing, involving as it often does the young and the active.

Numerous surgical techniques have been developed to treat these injuries, but none has yet been shown to be superior. One of the most widely employed and best-studied means of achieving cartilage repair in patients with discrete regions of chondral destruction in the knee is that of microfracture. Microfracture is an arthroscopic technique that involves penetrating the subchondral bone at the base of full-thickness articular cartilage defects, thus allowing marrow pluripotent stem cells to egress into the chondral defect, facilitating cartilage repair. However, doubts have been raised concerning the quality and durability of the microfracture-induced repair tissue. In recent years, autologous chondrocyte implantation (ACI) has emerged as the technique with the greatest potential for advancing the management of chondral injury. In this procedure, autologous chondrocytes are harvested from non-critical areas on the articular surface, then expanded through cell culture in the laboratory, before being implanted 4-6 weeks later into the chondral defect, using a 'patch' of adjacent periosteum for containment of the cells within the defect. There are several disadvantages to the ACI technique just described: it is a two-stage procedure, chondrocyte culture can be lengthy and expensive, and the periosteal patch used to contain the cells is associated with a significant risk of complications such as detachment and hypertrophy. 2nd generation ACI techniques have focused on addressing some of these problems by substituting the periosteum patch with artificial membranes that served as scaffolds for the cultured chondrocytes.

A novel technique has recently been developed that could prove to avoid some of the deficiencies of the ACI technique. The Cartilage Autograft Implantation System (CAIS) is a single-stage procedure in which cartilage is harvested from non-critical regions of articular cartilage, but then immediately morcellated and loaded onto a polymer membrane-scaffold, which is subsequently used to fill the chondral defect. The autograft-membrane composite is fixed to the defect with a biodegradable staple.

We aim to evaluate this new technique through a pilot clinical trial involving 36 patients randomized into microfracture and CAIS treatment arms (randomisation ratio 1:2), with a minimum follow-up of 1 year, using both clinical and radiological (magnetic resonance imaging) outcomes. If the results of this pilot trial are successful, we plan to expand the study by recruiting more patients to achieve a suitably-powered trial.

Primary hypothesis 1: That functional scores will increase by at least 0.5 SD over pre-operative values, by 1 year following the CAIS procedure

Primary hypothesis 2: That articular cartilage height will have a sustained increase of at least 2 mm at 1 year following the CAIS procedure

Primary hypothesis 3: That functional scores in the CAIS group will be equivalent or superior to those in the microfracture group

ELIGIBILITY:
Inclusion Criteria:

* Full-thickness articular cartilage defect on the femoral condyle or trochlea greater than 2 cm2 but less than 10 cm2 in total surface area, following debridement to healthy, stable tissue.
* Knee mechanical axis malalignment of not more than 3 degrees either varus or valgus from neutral.
* Patient is fit for surgery.

Exclusion Criteria:

* Multifocal disease
* Tibial plateau lesions
* Patella lesions
* Absent menisci or meniscal tears that are unstable and cannot be successfully debrided
* Non-intact cruciate and collateral ligaments
* Inflammatory or crystalline arthropathy
* Systemic medication or conditions likely to compromise chondrocyte cell proliferation and differentiation, e.g. Cushing's syndrome, chemotherapy
* Morbid obesity (more than 150% ideal body weight)

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
MR Observations of Cartilage Repair Tissue | 3 weeks post operative
  The MOCART (MR Observations of Cartilage Repair Tissue) scoring system, which has been well validated in studies of cartilage regeneration techniques, will be used to assess the cartilage repair response
MR Observations of Cartilage Repair Tissue | 6 months post-operative
  The MOCART (MR Observations of Cartilage Repair Tissue) scoring system, which has been well validated in studies of cartilage regeneration techniques, will be used to assess the cartilage repair response
MR Observations of Cartilage Repair Tissue | 1 year post-operative
  The MOCART (MR Observations of Cartilage Repair Tissue) scoring system, which has been well validated in studies of cartilage regeneration techniques, will be used to assess the cartilage repair response

SECONDARY OUTCOMES:
Assessment of whole leg mechanical alignment | 1 week prior to surgery
  Standard weight-bearing plain radiographs of the knee, as well as long leg standing films to assess mechanical alignment, will also be performed.
Assessment of whole leg mechanical alignment | 1 month post-operative
  Standard weight-bearing plain radiographs of the knee, as well as long leg standing films to assess mechanical alignment, will also be performed.
Assessment of whole leg mechanical alignment | 3 month post-operative
  Standard weight-bearing plain radiographs of the knee, as well as long leg standing films to assess mechanical alignment, will also be performed.
Assessment of whole leg mechanical alignment | 6 month post-operative
  Standard weight-bearing plain radiographs of the knee, as well as long leg standing films to assess mechanical alignment, will also be performed.
Assessment of whole leg mechanical alignment | 1 year post-operative
  Standard weight-bearing plain radiographs of the knee, as well as long leg standing films to assess mechanical alignment, will also be performed.
Clinical and functional evaluation using standardised and validated scoring system | 1 week prior to surgery
  Pre- and post-operative assessment (1,3,6 and 12 months) of the diseased knee will be performed using standardised, validated scoring systems: SF-36 (general health), KOOS and ICRS (disease-specific) scores
Clinical and functional evaluation using standardised and validated scoring system | 1 month post-operative
  Pre- and post-operative assessment (1,3,6 and 12 months) of the diseased knee will be performed using standardised, validated scoring systems: SF-36 (general health), KOOS and ICRS (disease-specific) scores
Clinical and functional evaluation using standardised and validated scoring system | 3 month post-operative
  Pre- and post-operative assessment (1,3,6 and 12 months) of the diseased knee will be performed using standardised, validated scoring systems: SF-36 (general health), KOOS and ICRS (disease-specific) scores
Clinical and functional evaluation using standardised and validated scoring system | 6 month post-operative
  Pre- and post-operative assessment (1,3,6 and 12 months) of the diseased knee will be performed using standardised, validated scoring systems: SF-36 (general health), KOOS and ICRS (disease-specific) scores
Clinical and functional evaluation using standardised and validated scoring system | 1 year post-operative
  Pre- and post-operative assessment (1,3,6 and 12 months) of the diseased knee will be performed using standardised, validated scoring systems: SF-36 (general health), KOOS and ICRS (disease-specific) scores

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Lu Chia, PhD, MBBS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore